CLINICAL TRIAL: NCT01371175
Title: A Randomized, Placebo-Controlled, Dosage-Escalating Phase 2A Study, Double-Blinded With Respect to Assignment to Either Vaccine or Placebo, to Evaluate the Safety and Immunogenicity of a DNA HIV-1 Vaccine Administered Intramuscularly Followed by an MVA HIV-1 Vaccine Administered at Three Different Dosage Levels and by Three Different Routes to HIV-Uninfected, Healthy, Volunteers.
Brief Title: A Phase IIA Trial to Evaluate the Safety and Immunogenicity of a DNA HIV-1 Vaccine Followed by an MVA HIV-1 Vaccine in HIV-uninfected Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: Medical Research Council-Oxford (Unknown); University of Nairobi (Other)
Responsible Party: Patricia Fast, MD, PhD. Chief Medical Officer, International AIDS Vaccine Initiative
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IAVI 010
Record Dates: First submitted 2011-05-31; First posted 2011-06-10 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Group A (Experimental): DNA or Placebo delivered intramuscularly at Months 0 and 1 followed by MVA or Placebo at Months 5 and 8 delivered subcutaneously. Vaccine:Placebo =12/3
  Interventions: Biological: DNA.HIVA; Biological: MVA.HIVA
- Group B (Experimental): DNA or Placebo delivered intramuscularly at Months 0 and 1 followed by MVA or Placebo at Months 5 and 8 delivered intramuscularly. Vaccine:Placebo =12/3
  Interventions: Biological: DNA.HIVA; Biological: MVA.HIVA
- Group C (Experimental): DNA or Placebo delivered intramuscularly at Months 0 and 1 followed by MVA or Placebo at Months 5 and 8 delivered intradermally. Vaccine:Placebo =18/3
  Interventions: Biological: DNA.HIVA; Biological: MVA.HIVA
- Group D (Experimental): DNA or Placebo delivered intramuscularly at Months 0 and 1 followed by MVA or Placebo at Months 5 and 8 delivered subcutaneously. Vaccine:Placebo =12/3
  Interventions: Biological: DNA.HIVA; Biological: MVA.HIVA
- Group E (Experimental): DNA or Placebo delivered intramuscularly at Months 0 and 1 followed by MVA or Placebo at Months 5 and 8 delivered intramuscularly. Vaccine:Placebo =12/3
  Interventions: Biological: DNA.HIVA; Biological: MVA.HIVA
- Group F (Experimental): DNA or Placebo delivered intramuscularly at Months 0 and 1 followed by MVA or Placebo at Months 5 and 8 delivered subcutaneously. Vaccine:Placebo =12/3
  Interventions: Biological: DNA.HIVA; Biological: MVA.HIVA
- Group G (Experimental): DNA or Placebo delivered intramuscularly at Months 0 and 1 followed by MVA or Placebo at Months 5 and 8 delivered intramuscularly. Vaccine:Placebo =12/3
  Interventions: Biological: DNA.HIVA
- Groups C2/D2/E2 (Subgroups of C,D,E) (Experimental): DNA or Placebo delivered intramuscularly at Months 0 and 1 followed by MVA or Placebo at Months 5 and Month 12+ (volunteers offered second MVA/placebo more than 12 months (late boost) after their enrollment into their original treatment assignment) delivered ID, SC, or IM according to original randomization. Vaccine:Placebo = blinded ratio, maximum in C2/D2/E2 = 16.
  Interventions: Biological: DNA.HIVA; Biological: MVA.HIVA
- Group F2/G2 (Subgroup of F and G) (Experimental): DNA or Placebo delivered intramuscularly at Months 0 and 1 followed by MVA or Placebo at Months 5 and Month 12+ (volunteers offered second MVA/placebo more than 12 months (late boost) after their enrollment into their original treatment assignment) delivered either SC or IM according to original randomization. Vaccine:Placebo = blinded ratio, maximum in F/G= 29.
  Interventions: Biological: DNA.HIVA; Biological: MVA.HIVA

INTERVENTIONS:
Biological: DNA.HIVA — 0.5mg DNA.HIVA or placebo
Biological: MVA.HIVA — 5x10^6 pfu MVA or placebo
  Arms: Group A; Group B
Biological: MVA.HIVA — 5x10^7 pfu MVA or placebo
  Arms: Group C; Group D; Group E; Groups C2/D2/E2 (Subgroups of C,D,E)
Biological: MVA.HIVA — 2.5x10^8 pfu MVA or placebo
  Arms: Group E; Group F; Group F2/G2 (Subgroup of F and G)

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of plasmid DNA and recombinant MVA (Modified Vaccinia Virus Ankara) in a prime-boost regimen.

Approximately 111 volunteers (90 vaccine recipients/21 placebo recipients) will be enrolled at two sites. Approximately 56 volunteers will be enrolled at each site. An over-enrolment of up to 10% (approximately 10 additional volunteers) will be permitted in the study.

ELIGIBILITY:
Inclusion Criteria

1. Healthy males and females;
2. Age at least 18 years on the day of screening and no greater than 60 years on the day of enrolment;
3. Available for follow up for the planned duration of the study (screening plus 18 months);
4. Able to give written informed consent;
5. Does not engage in risk behaviour as defined by the protocol, willing to undergo HIV testing and receive results;
6. If sexually active female, using an effective method of contraception (combined oral contraceptive pill; injectable contraceptive; IUCD; condoms; anatomical sterility in self or partner) from screening until at least 4 months after last vaccination and willing to undergo urine pregnancy tests at screening and prior to each vaccination and 4 months after the last vaccination;
7. If sexually active male, willing to use an effective method of contraception (such as condoms) from screening until 4 months after the last vaccination.

Exclusion Criteria:

1. Clinically relevant abnormality on history or examination including history of immunodeficiency or use of systemic corticosteroids, immunosuppressive, antiviral, anticancer, or other medications considered significant by the designated trial physician in last 6 months;
2. Presence of any chronic condition;
3. Any of the following abnormal laboratory parameters that are moderate, severe, or very severe: haematology (haemoglobin, absolute neutrophil count absolute lymphocyte count , absolute CD4 count, platelets); urinalysis, biochemistries (total bilirubin, creatinine, AST, ALT). Volunteers with mild laboratory abnormalities which are judged by the principal investigator or designee to be not clinically significant may be enrolled.
4. If female, pregnant or planning a pregnancy within 4 months after last vaccination or lactating;
5. Receipt of live attenuated vaccine within 60 days or other vaccine within 14 days of enrolment;
6. Receipt of blood transfusion or blood products 6 months prior to enrolment;
7. Participation in another clinical trial of an investigational product currently or within last 12 weeks or expected participation during this study;
8. History of severe local or general reaction to vaccination or history of allergic reactions;
9. History of grand-mal epilepsy, or currently taking anti-epileptics;
10. Confirmed HIV-1 or HIV-2 seropositive;
11. Positive for hepatitis B (surface antigen) or confirmed diagnosis of active syphilis at the time of enrolment (RPR positive and TPHA positive or equivalent), positive for hepatitis C antibodies;
12. Unlikely to comply with protocol. Prior receipt of smallpox vaccination should be documented, but will not be an exclusion criterion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2003-04; Primary Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Safety (local and systemic reactogenicity signs and symptoms, laboratory measures, and adverse events) | 18 months

SECONDARY OUTCOMES:
Immunogenicity: Proportion of volunteers with HIV-1 specific T-cell responses by ELISPOT assay. | Day 0, Month 1, Month 2, Month 5, Month 6, Month 8, Month 9, Month 12, Month 18

CONTACTS AND LOCATIONS:
Overall Officials: Barry S. Peters, MD, Principal Investigator — Guys and St. Thomas' Hospital; Walter Jaoko, Principal Investigator — KAVI (Kenya AIDS Vaccine Initiative)
Locations (2):
- KAVI (Kenya AIDS Vaccine Initiative), Nairobi, Kenya
- Guys and St. Thomas' Hospital, London, United Kingdom

REFERENCES:
- See also: International AIDS Vaccine Initiative — http://www.iavi.org